CLINICAL TRIAL: NCT02585661
Title: Iron Bioavailability From Fortified Dairy Product in Healthy Women
Brief Title: Iron Bioavailability From Dairy Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15.06.MET
Record Dates: First submitted 2015-10-16; First posted 2015-10-23 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dairy product + Salt 1 (Active Comparator): Dairy product fortified with enriched Fe-54 salt (1)
  Interventions: Dietary Supplement: Dairy product fortified with enriched Fe-54 salt (1)
- Dairy product + Salt 2 (Experimental): Dairy product fortified with enriched Fe-57 salt (2)
  Interventions: Dietary Supplement: Dairy product fortified with enriched Fe-57 salt (2)

INTERVENTIONS:
Dietary Supplement: Dairy product fortified with enriched Fe-54 salt (1) — 2.5mg of Fe per 100g of product
  Arms: Dairy product + Salt 1
Dietary Supplement: Dairy product fortified with enriched Fe-57 salt (2) — 2.5mg of Fe per 100g of product
  Arms: Dairy product + Salt 2

SUMMARY:
Determination of fractional iron absorption from dairy product fortified with 2 labelled iron compounds

DETAILED DESCRIPTION:
This single center trial will be double-blind, controlled randomized with a crossover trial. One group (n=10) will start the study with the consumption of a Fe-54 salt fortified dairy product, while the other group will start the study with the consumption of Fe-57 salt fortified dairy product. The day after, in a cross over design, subjects will be administered the alternative test product. A blood sampling will be performed 14 days after the last stable isotope administration to allow the measurement of Fe stable isotope ratios and the calculation of Fe absorption. The duration of the trial will be 16 days in total.

The total sample size is 20 enrolled subjects. Patients will be healthy females aged 18-40 years old

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years old,
* Healthy, based on the medical screening visit including a blood formula and biochemistry,
* Normal BMI for age (18.5-25.0),
* Weight less than 65 kg,
* Having obtained informed consent prior trial entry.

Exclusion Criteria:

* Anemia or polycythemia respectively evidenced,
* Significant blood losses over the past 6 months,
* Plasma ferritin out of 8-50 ug/L range.
* Any infectious and inflammatory disease in the past four weeks,
* Relevant digestive (intestinal, gastric, hepatic or pancreatic), renal, metabolic disease,
* Known food allergy,
* Pregnancy (anamnesis) and/or lactation,
* History of cancer within the past year,
* Significant weight loss during the last 3 months (5% and more),
* medication or supplement which may impact red cells count, Hb or Ht
* Fe supplementation or perfusion in the last three months,
* Smokers (>5 cigarettes),
* Have a high alcohol consumption (more than 2 drinks/day),
* Consumption of illicit drugs anamnesis only,
* Subject having a hierarchical link with the Investigator or co-investigators,
* Subject who cannot be expected to comply with treatment or study procedure,
* participating or having participated in another clinical trial during the past month prior to the beginning of this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | 14 days after the last stable isotope administration
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes

SECONDARY OUTCOMES:
Measurement of plasma ferritin as biomarker of Fe status | On the 1st day of the stable isotope administration
  The plasma ferritin will be measured before the administration of test meal including iron isotopes

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, Principal Investigator — Metabolic Unit - Nestec
Locations (1):
- Metabolic Unit, Clinical Development Unit, Nestec, Lausanne, Switzerland